CLINICAL TRIAL: NCT01149408
Title: A Pilot Study of Decitabine Maintenance in Elderly Acute Myeloid Leukemia Patients Who Can Tolerate Aggressive Therapy
Brief Title: Decitabine Maintenance in Elderly Acute Myeloid Leukemia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI42887
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Acute Myeloid Leukemia; AML
Keywords: AML; Decitabine; Acute Myeloid Leukemia; Elderly Patients; Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Drug: Decitabine (Dacogen)

INTERVENTIONS:
Drug: Decitabine (Dacogen) — Decitabine; 20 mg/m2; 1 hour intravenous infusion; 1 -3 days (will be given on a 28-day cycle for up to 18 months)
  Other Names: Dacogen (NDA 021790)

SUMMARY:
The study aims at determining the feasibility of using maintenance Decitabine therapy following remission induction and consolidation in elderly Acute Myeloid Leukemia patients who are fit for aggressive therapy.

Primary: Safety and tolerability of the decitabine regimen in the post remission state.

Secondary:

1. Disease-free survival - To determine the one-year disease-free survival in elderly patients with acute myeloid leukemia (AML) in complete remission treated with Decitabine as post-consolidation maintenance therapy.
2. Overall survival

DETAILED DESCRIPTION:
The median age of patients with AML at presentation is between 65 to 70 years (Peterson 1977, Brincker 1985, Baudard 1994) and the incidence of AML increases with advancing age (Wingo 1995). Given this, increased attention should be focused on adult patients 60 years or older with this disease. Treatment strategies in younger patients are well established however therapy in the elderly deserves particular thought (Foon 1981, Sebban 1998, Lowenberg 1998). Also progress in the treatment of AML in the elderly population is not near progress that has been made in the treatment of the younger population (Stone 2002, Kantarjian 2006). Poor tolerability and questionable treatment benefit have left older adult patients with AML often without effective treatment options or with best supportive care. According to Medicare records, only 30% of a cohort of 2657 AML patients older than 65 years were provided chemotherapy treatment (44% in patients 65 to 74 years, 24% in patients 75 to 84, and 6% in patients 85 and above). The mortality was 86% at 1 year and 94% at 2 years following the diagnosis. The overall survival in this cohort was only 2 months (Menzin 2002). The study could not distinguish between intensive induction chemotherapy and palliative therapy.

Despite modest improvements in outcomes for younger patients with AML, adults over 55 years of age (the majority of patients with AML) continue to do poorly (Tallman 2005).

In patients over 60 years response rates have ranged from 40% to 55% and in patients over 70 years have ranged from 24% to 33% (Buchner 2009, Estey 2007, Lowenberg 1998, Rowe 2004). Patient and leukemia related factors could explain the poor result of older patients with AML (Harry 2007, Gupta 2005). Also in patients over 60, with adverse cytogenetics the response rates range from 26% to 34%; with antecedent hematologic disorder they range between 28% and 46%; and with Eastern Cooperative Oncology Group (ECOG) performance status (PS) 2 it is around 26%. (Grimwade 2001, Rowe 2004, Appelbaum 2006).

For the past several decades, standard induction chemotherapy for acute myeloid leukemia (AML) has consisted of the "7+3" regimen of cytarabine plus an anthracycline. Standard consolidation chemotherapy has consisted of high dose cytarabine for 3-4 cycles. Few trials have randomized older patients with AML to receive standard remission induction (i.e., anthracycline-containing) chemotherapy versus either palliative therapy or less intensive chemotherapy. The median survival of older adults with AML treated with cytarabine plus an anthracycline on the "7+3" schedule is 8 to 12 months (Estey 2007, Rowe 2004). Less than 10% of patients remain in remission for more than 3 years. (Lowenberg 1998, Godwin 2003, Roboz 2007).

The European Organization for the Research and Treatment of Cancer (EORTC) conducted a trial on 60 patients and randomized them to intensive chemotherapy (daunorubicin 30 mg/m2/day intravenously [IV] for 3 days, vincristine 1 mg/m2/day IV on Day 2, cytarabine 100 mg/m2/day IV for 7 days with 50 mg/m2/day IV bolus every 12 hours for 7 days) or a "watch and wait" approach (supportive care alone with hydroxyurea 3 g PO on Days 1 and 4 and LDAC (subcutaneous cytarabine) 100 mg/m2 every 12 hours SC on Days 2, 3, 5, and 6 administered only when leukemia-related symptoms occurred). All patients were more than 65 years old, but had to have preserved organ function and performance status. The patients who received induction chemotherapy had a higher complete remission (CR) rate (58% vs. 0%), lower incidence of early mortality (3/31 vs. 18/29 patients), longer median survival (21 weeks vs. 11 weeks) and greater chance of survival at 2.5 years (17% vs. 0%). The median duration of hospitalization did not statistically differ between the two groups.

In the study performed by Tilly et al (Tilly 1990) in patients >65 years old, 87 patients were randomized to receive either LDAC 10 mg/m2 SC every 12 hours for 21 days or standard chemotherapy induction with rubidazone (a daunorubicin-derived agent) 100 mg/m2 IV for 4 days plus cytarabine 200 mg/m2 IV for 7 days. The combination chemotherapy arm was associated with a 31% early death rate compared with10% in the lower dose arm. There was a higher CR rate in the rubidazone/cytarabine arm (52% versus 32%), but only a trend toward improved survival favoring this arm (12.8 months versus 8.8 months) was reported.

Repetitive cycles of high dose Cytarabine (HiDAC- 3 g/m2 ARA-C twice a day on days 1, 3, 5) is an effective consolidation regimen for AML patients based on the CALGB in 1994 (Mayer 1994). In patients younger than 60, this protocol produced a high rate of continuous CR. However in patients older than 60, a high rate of neurotoxicity was reported using this regimen (Mayer 1994). A follow up study modified this protocol by using Intermediate Dose Cytarabine (IDAC) (1 g/m2 ARA-C twice a day on days 1, 3, 5) and applied the regimen to a group of elderly patients (≥60 years) with de novo AML. This protocol (IDAC) was found to be an effective and well-tolerated consolidation regimen for elderly patients (Sperr 2004). Based on this study the median overall survival, disease-free survival, and continuous CR were 10.6, 15.5, and 15.9 months, respectively (Sperr 2004).

Thus, from the data obtained in these studies, chemotherapy in some form is superior to best supportive care alone or best supportive care with chemotherapy initiated after evidence of disease progression. However no single treatment approach appears adequate and can be considered the standard of care for elderly AML patients. Thus, improved treatment strategies and more suitable chemotherapy regimens are needed (Harry 2007). Additionally, it is not clear how best to administer chemotherapy with currently available drugs, taking into account induction and consolidation treatments.

Several different categories of new therapies are under development, including multidrug resistance (MDR) reversal agents, immunomodulatory therapies, and signal transduction targeting. Table 1 shows examples of targets and agents developed and being developed. Given the lack of standards in the treatment of elderly AML, of the use of these newer agents in treating AML is justified.

Table 1: Targets for New Agents for Acute Myelogenous Leukemia (Medscape.com) Targets Agents CD33 Gemtuzumab ozogamicin CD45 131I-anti-CD45 MDR1/Pgp Cyclosporine, PSC-833 Angiogenesis and/or VEGF Thalidomide, SU-5416, bevacizumab antibodies Hypermethylated chromatin Decitabine Histone deacetylase Phenylbutyrate trichostatin A, trapoxin Bcl-2 Bcl-2 antisense S-phase checkpoint UCN-01 20S proteasome PS-341 Tyrosine kinase (c-kit receptor) STI-571 Flt-3 kinase CEP-701 Farnesyl transferase BMS-214662, R115777

A sizeable percentage of older adults attain a complete remission with induction chemotherapy, but almost all of these patients will relapse within a median of four to eight months unless given additional cytotoxic therapy (Cassileth 1999). Even with post-remission therapy, relapses are common. Furthermore, post-remission therapy in older adults is complicated by high rates of treatment related toxicity.

To address the problem of post-remission therapy, the Nordic MDS group performed a phase II multicenter study, which studied long-term maintenance with azacitidine. They studied patients with high-risk MDS and AML arising from MDS. The mean age of the group was 68 years. Patients who achieved CR after induction received low dose azacitidine sq 5 out of 28 days until relapse. They noted a median CR duration of 13.5 months and noted very mild side effects (Grovdal 2008).

In another phase II trial Decitabine was used for untreated AML patients older than 60 who were not candidates for intensive chemotherapy (or who refused it). PS was ECOG <3. All pts received induction with Decitabine at 20mg/m2 IV on days 1-10 of a 4 week cycles. Patients with persistent AML at the end of a cycle received a repeat of the 10 day course, but responding patients received maintenance with shortened courses of 3-5 days depending on the degree and duration of neutropenia. Forty two percent of patients achieved CR. Median OS has not yet been reached; median f/u of 19 surviving patients was 8 months. The median number of cycles received till the date of publication was five (Blum 2009).

One retrospective study studied 141 elderly AML patients in first CR after 7+3 induction chemotherapy. In patients aged 60-70 year, consolidation ± maintenance therapy improved outcomes (DFS and OS). In patients older than 70 and with WBC < 30 x109/l maintenance therapy without consolidation improved outcomes. In patients older than 70 and with WBC < 30 x 109/l consolidation therapy worsened outcomes. In patients older than 70 and with WBC > 30 x 109/l, both consolidation and/or maintenance therapy did not improve outcomes (Corre 2005).

The purpose of this study is to determine whether it is feasible to use maintenance treatment (prolonged treatment over several months) with Decitabine in elderly patients with AML after they have obtained a remission with standard chemotherapy. The study also aims at obtaining preliminary results on whether this approach prolongs the period of remission after standard chemotherapy. The study group will include elderly (≥60 years of age), Acute Myeloid Leukemia (AML) patients who can tolerate an aggressive therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AML (excluding Acute Promyelocytic Leukemia) according to the WHO classification, including de novo and secondary AML. Patient must be in complete remission after 1 cycle of induction therapy consisting of cytarabine (100 mg/m2 as a 24 hour infusion for 7 consecutive days) and idarubicin (12 mg/m2 as a slow intravenous push daily for 3 days), and 2 cycles of consolidation therapy (each consisting of cytarabine at a dose of 1 g/m2 given intravenously over 3 hours every 12 hours on days 1,3,and 5).
2. Patients who maintain morphologic complete remission as documented by a bone marrow aspirate/biopsy after consolidation therapy will be eligible to receive Decitabine maintenance therapy. Maintenance therapy should be started as soon as feasible after recovery from the last consolidation cycle but no sooner than 29 days after start of the last consolidation cycle and no later than 60 days after recovery from the last cycle of consolidation therapy.
3. Age ≥ 60 years
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. Informed consent, personally signed and dated to participate in the study
6. Be able to comply with study procedures and follow-up examinations
7. Be non-fertile or agree to use birth control during the study through the end of last treatment visit
8. Adequate renal and hepatic function as indicated by all of the following: Total bilirubin ≤ 1.5 institutional Upper Limit of Normal (ULN); and Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 ULN; and Serum creatinine ≤ 1.5 mg/dL
9. Adequate cardiac function as measured by at least 1 of the following: Left ventricular ejection fraction (LVEF) ≥ 50% on multigated acquisition (MUGA) scan, similar radionuclide angiographic scan, or echocardiogram

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL, WHO classification of APL with t(15;17)(q22;q12)
2. Prior diagnosis and treatment for AML, including hematopoietic stem cell transplant (HSCT)
3. Previous therapy with a hypomethylating agent including decitabine or azacitidine (i.e. for an antecedent myelodysplastic syndrome)
4. Any prior therapy for AML except for hydroxyurea for the control of blood counts
5. Psychiatric disorders that would interfere with consent, study participation, or follow-up
6. Cardiac Disease: Heart failure NYHA class 3 or 4; unstable coronary artery disease (MI more than 6 months prior to study entry is permitted); serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
7. Chronically impaired renal function (creatinine clearance < 30 ml / min)
8. Inadequate liver function (ALT and AST ≥ 2.5 x ULN) if not caused by leukemic infiltration
9. Total bilirubin ≥ 1.5 x ULN if not caused by leukemic infiltration
10. Known HIV and/or hepatitis C infection
11. Evidence or history of severe non-leukemia associated bleeding diathesis or coagulopathy
12. Evidence or recent history of CNS disease, including primary or metastatic brain tumors, seizure disorders
13. Clinical evidence suggestive of central nervous system (CNS) involvement with leukemia unless a lumbar puncture confirms the absence of leukemic blasts in the cerebrospinal fluid (CSF)
14. Any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo therapy on this protocol
15. Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
16. Diagnosis of another malignancy, unless the patient has been disease-free for at least 5 years following the completion of curative intent therapy with the following exceptions: Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed. Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed
17. History of organ allograft
18. Any severe concomitant condition, which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol
19. Patients who have an indication for and can undergo a non-myeloablative transplant procedure

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Primary: Safety and tolerability of the decitabine regimen in the post remission state. | 18 mos on treatment and one year followup thereafter
  Patient will come to the infusion center for a one-hour infusion on three (3) consecutive days during a 28-day cycle. The 28-day cycle will be repeated for up to 18 months if tolerated or there is no evidence of loss of remission. Patient will receive maintenance therapy with the study drug Decitabine.
  The Long-Term Follow-Up Schedule begins from the end of treatment. All patients who receive at least one dose of study drug will be followed for a minimum of one year. The maximum follow-up for all patients will be 5 years from the date of last enrolled patient.

SECONDARY OUTCOMES:
1- Disease-free survival - | One Year
  To determine the one-year disease-free survival in elderly patients with acute myeloid leukemia (AML) in complete remission treated with Dectiabine as post-consolidation maintenance therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Shami, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah, United States